CLINICAL TRIAL: NCT05888415
Title: WELL-being Improvement Following Sophrology Practice
Acronym: SoWell-Learn
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Responsible Party: Sponsor
Other Study IDs: RNI 2022 DUTHEIL 2
Record Dates: First submitted 2023-04-25; First posted 2023-06-05 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Well-being

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- sophrology practitioners: Practice sophrology - no intervention
- non practitioners: Do not practice sophrology - no intervention

SUMMARY:
Stress and psychosocial risks are a major public health problem.Sophrology is a psycho-corporal method exclusively verbal and non-tactile used as a therapeutic technique. It combines a set of techniques that will act both on the body and on the mind through breathing exercises, muscle relaxation and mental imagery (or visualization). It allows to find a state of well-being and to activate all physical and psychological potential in order to acquire a better knowledge of oneself. Sophrology demonstrated some benefits on symptoms of patients. However, these approaches have never been evaluated with a prolonged follow-up of several months, with biological measures or with adjustments according to the levels of mastery of sophrology. This project proposes to evaluate the effects of sophrology practice. The investigators aim to evaluate both subjective and objective measures of stress.

DETAILED DESCRIPTION:
Those interested in participating in the study will contact the investigators via the email address provided on the flyer. A clinical research associate will contact them and give them an appointment at the Institute of Occupational Medicine, Faculty of Medicine, 28 place Henri Dunant, 63000 Clermont-Ferrand, in order to provide them with informed information and respond to their their questions.

If participants agree to participate, the clinical research associate will provide them with the saliva collection kit with instructions for use and a Redcap® link to inform their commitment, and complete an inclusion questionnaire and the first main questionnaire. Then, the participants will receive the questionnaire directly by email for the following fillings.

When accessing Redcap®, a brief description of the study will again be provided. We will ask the participant to commit to their group's inclusion criteria by checking a box. The non-opposition will be collected by clicking on "envoyer" at the end of the information letter. The following sentence will be indicated "In the case of an agreement please click on the button "envoyer".

After collection of the non-opposition, participant will have to completed a short inclusion questionnaire composed of:

* Initials for create an ID
* Sociodemographic variables: gender, age, marital status, children, occupation, and recent stressful event.
* Group : " pratiquant " or " non pratiquant ". For those practicing sophrology: type of practice and number of years of practice
* Realization of another wellness practice
* Email address to be able to receive the questionnaires each month by automatic sending. In order to guarantee anonymity, the email address of the participants will not be accessible to the investigators / collaborators of the study. They will thus be contacted by email directly by REDCap® for the questionnaire filling (identical questionnaire each month during 6 months).

The self-administered main questionnaire will be composed of:

* Information about saliva sampling: Date and time of collection, Time of awakening on day of collection, Eppendorf number
* Visual analog scales assessing the perceived stress, anxiety, sleep quality, fatigue, time judgment and emotions on a horizontal, non-calibrated line of 100 mm, ranging from very low (0) to very high (100).
* Lifestyle variables: treatment, physical activity, addiction (alcohol, cannabis, and tobacco), coffee/tea and food intake.
* Sophrology practice: Number of sessions per week, type of practice, stress before and after the last sophrology session, realization of another wellness practice

Furthermore, each participant will do a self-collection of saliva the first week of each month, upon waking up, on a day of the week chosen by the participant as being as reproducible as possible. Participants will have to keep the samples in their freezer and bring them back to us in an ice pack at the end of the 6 months. For this purpose, in the last questionnaire, we will display a window asking them to contact us to organise the return of their saliva samples.

ELIGIBILITY:
Inclusion criteria

For both groups (sophro-practitioners vs. non-practitioners), being able to give informed consent to participate in the research. Commit to respecting the inclusion criteria of their group.

* For sophro-practitioners:

  * practice at least once a week,
  * practice vertically following the dynamic relaxation method.
* For non-practitioners, do not practice sophrology during the follow-up. If the participant changes his mind, he will be asked to inform the investigator.

Exclusion Criteria:

* Protected persons (minors, pregnant women, breastfeeding women, guardianship, curatorship, deprived of freedoms, safeguard of justice)
* Refusal to participate

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The study is composed of a group of people practicing sophrology and a group of people who do not practice it
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-06-19 (Actual); Primary Completion 2023-12-27 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
DHEAS | Baseline
  Stress measure objectively using dheas measured in pg/ml
Cortisol | Baseline
  Stress measure objectively using cortisol measured in µg/dl
Leptine | Baseline
  Stress measure objectively using leptin measured in ng/ml
Ghrelin | Baseline
  Stress measure objectively using ghrelin measured in pg/ml
DHEAS | month 1
  Stress measure objectively using dheas measured in pg/ml
Cortisol | month 1
  Stress measure objectively using cortisol measured in µg/dl
Leptin | month 1
  Stress measure objectively using leptin measured in ng/ml
Ghrelin | month 1
  Stress measure objectively using ghrelin measured in pg/ml
DHEAS | month 2
  Stress measure objectively using dheas measured in pg/ml
Cortisol | month 2
  Stress measure objectively using cortisol measured in µg/dl
Leptin | month 2
  Stress measure objectively using leptin measured in ng/ml
Ghrelin | month 2
  Stress measure objectively using ghrelin measured in pg/ml
DHEAS | month 3
  Stress measure objectively using dheas measured in pg/ml
Cortisol | month 3
  Stress measure objectively using cortisol measured in µg/dl
Leptin | month 3
  Stress measure objectively using leptin measured in ng/ml
Ghrelin | month 3
  Stress measure objectively using ghrelin measured in pg/ml
DHEAS | month 4
  Stress measure objectively using dheas measured in pg/ml
Cortisol | month 4
  Stress measure objectively using cortisol measured in µg/dl
Leptin | month 4
  Stress measure objectively using leptin measured in ng/ml
Ghrelin | month 4
  Stress measure objectively using ghrelin measured in pg/ml
DHEAS | month 5
  Stress measure objectively using dheas measured in pg/ml
Cortisol | month 5
  Stress measure objectively using cortisol measured in µg/dl
Leptin | month 5
  Stress measure objectively using leptin measured in ng/ml
Ghrelin | month 5
  Stress measure objectively using ghrelin measured in pg/ml
DHEAS | month 6
  Stress measure objectively using dheas measured in pg/ml
Cortisol | month 6
  Stress measure objectively using cortisol measured in µg/dl
Leptin | month 6
  Stress measure objectively using leptin measured in ng/ml
Ghrelin | month 6
  Stress measure objectively using ghrelin measured in pg/ml
Subjective stress | Baseline
  stress measure subjectively using a visual analogue scale ranging from 0 (minimum) to 100 (maximum)
Subjective stress | Month 1
  stress measure subjectively using a visual analogue scale ranging from 0 (minimum) to 100 (maximum)
Subjective stress | Month 2
  stress measure subjectively using a visual analogue scale ranging from 0 (minimum) to 100 (maximum)
Subjective stress | Month 3
  stress measure subjectively using a visual analogue scale ranging from 0 (minimum) to 100 (maximum)
Subjective stress | Month 4
  stress measure subjectively using a visual analogue scale ranging from 0 (minimum) to 100 (maximum)
Subjective stress | Month 5
  stress measure subjectively using a visual analogue scale ranging from 0 (minimum) to 100 (maximum)
Subjective stress | Month 6
  stress measure subjectively using a visual analogue scale ranging from 0 (minimum) to 100 (maximum)

SECONDARY OUTCOMES:
Sociodemographic | once at baseline
  gender, age, marital status, children, occupation, and recent stressful event
Sophrology practice | once at baseline
  Type of sophrology practice using a multiple-choice question
Drug treatment | Baseline
  Multiple-choice question: "Do you take long-term medication? No treatment, Psychotropics, Sleeping pills, Antihypertensives, etc."
Drug treatment | Month 1
  Multiple-choice question: "Do you take long-term medication? No treatment, Psychotropics, Sleeping pills, Antihypertensives, etc."
Drug treatment | Month 2
  Multiple-choice question: "Do you take long-term medication? No treatment, Psychotropics, Sleeping pills, Antihypertensives, etc."
Drug treatment | Month 3
  Multiple-choice question: "Do you take long-term medication? No treatment, Psychotropics, Sleeping pills, Antihypertensives, etc." If yes, "type of treatment" and "number of tablets per day"
Drug treatment | Month 4
  Multiple-choice question: "Do you take long-term medication? No treatment, Psychotropics, Sleeping pills, Antihypertensives, etc."
Drug treatment | Month 5
  Multiple-choice question: "Do you take long-term medication? No treatment, Psychotropics, Sleeping pills, Antihypertensives, etc."
Drug treatment | Month 6
  Multiple-choice question: "Do you take long-term medication? No treatment, Psychotropics, Sleeping pills, Antihypertensives, etc."
Tobacco consumption | Baseline
  Average number of cigarettes per day over the past month
Coffee consumption | Baseline
  Average number of cups of coffee per day over the past month
Tea consumption | Baseline
  Average number of cups of tea per day over the past month
Tobacco consumption | Month 1
  Average number of cigarettes per day over the past month
Coffee consumption | Month 1
  Average number of cups of coffee per day over the past month
Tea consumption | Month 1
  Average number of cups of tea per day over the past month
Tobacco consumption | Month 2
  Average number of cigarettes per day over the past month
Coffee consumption | Month 2
  Average number of cups of coffee per day over the past month
Tea consumption | Month 2
  Average number of cups of tea per day over the past month
Tobacco consumption | Month 3
  Average number of cigarettes per day over the past month
Coffee consumption | Month 3
  Average number of cups of coffee per day over the past month
Tea consumption | Month 3
  Average number of cups of tea per day over the past month
Tobacco consumption | Month 4
  Average number of cigarettes per day over the past month
Coffee consumption | Month 4
  Average number of cups of coffee per day over the past month
Tea consumption | Month 4
  Average number of cups of tea per day over the past month
Tobacco consumption | Month 5
  Average number of cigarettes per day over the past month
Coffee consumption | Month 5
  Average number of cups of coffee per day over the past month
Tea consumption | Month 5
  Average number of cups of tea per day over the past month
Tobacco consumption | Month 6
  Average number of cigarettes per day over the past month
Coffee consumption | Month 6
  Average number of cups of coffee per day over the past month
Tea consumption | Month 6
  Average number of cups of tea per day over the past month
Alcohol consumption | Baseline
  Average number of alcoholic drinks per week
Cannabis consumption | Baseline
  Average number of cannabis joints per week
Alcohol consumption | Month 1
  Average number of alcoholic drinks per week
Cannabis consumption | Month 1
  Average number of cannabis joints per week
Alcohol consumption | Month 2
  Average number of alcoholic drinks per week
Cannabis consumption | Month 2
  Average number of cannabis joints per week
Alcohol consumption | Month 3
  Average number of alcoholic drinks per week
Cannabis consumption | Month 3
  Average number of cannabis joints per week
Alcohol consumption | Month 4
  Average number of alcoholic drinks per week
Cannabis consumption | Month 4
  Average number of cannabis joints per week
Alcohol consumption | Month 5
  Average number of alcoholic drinks per week
Cannabis consumption | Month 5
  Average number of cannabis joints per week
Alcohol consumption | Month 6
  Average number of alcoholic drinks per week
Cannabis consumption | Month 6
  Average number of cannabis joints per week
Food consumption | Baseline
  Average food consumption in the last month
Food consumption | Month 1
  Average food consumption in the last month
Food consumption | Month 2
  Average food consumption in the last month
Food consumption | Month 3
  Average food consumption in the last month
Food consumption | Month 4
  Average food consumption in the last month
Food consumption | Month 5
  Average food consumption in the last month
Food consumption | Month 6
  Average food consumption in the last month
Physical activity | Baseline
  Average number of hours of physical activity per week over the past month
Physical activity | Month 1
  Average number of hours of physical activity per week over the past month
Physical activity | Month 2
  Average number of hours of physical activity per week over the past month
Physical activity | Month 3
  Average number of hours of physical activity per week over the past month
Physical activity | Month 4
  Average number of hours of physical activity per week over the past month
Physical activity | Month 5
  Average number of hours of physical activity per week over the past month
Physical activity | Month 6
  Average number of hours of physical activity per week over the past month
Well-being | Baseline
  Well-being measured using a visual analogue scale ranging from 0 (minimum) to 100 (maximum)
Well-being | Month 1
  Well-being measured using a visual analogue scale ranging from 0 (minimum) to 100 (maximum)
Well-being | Month 2
  Well-being measured using a visual analogue scale ranging from 0 (minimum) to 100 (maximum)
Well-being | Month 3
  Well-being measured using a visual analogue scale ranging from 0 (minimum) to 100 (maximum)
Well-being | Month 4
  Well-being measured using a visual analogue scale ranging from 0 (minimum) to 100 (maximum)
Well-being | Month 5
  Well-being measured using a visual analogue scale ranging from 0 (minimum) to 100 (maximum)
Well-being | Month 6
  Well-being measured using a visual analogue scale ranging from 0 (minimum) to 100 (maximum)

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Clemront-Ferrand, Clermont-Ferrand, France

IPD SHARING:
Plan to Share IPD: No